CLINICAL TRIAL: NCT04347473
Title: A Single Center Study to Evaluate the Effectiveness and Safety of ILUMYA in Combination With HALOG Ointment 0.1% for the Treatment of Moderate to Severe Plaque Psoriasis.
Brief Title: ILUMYA in Combination With HALOG Ointment 0.1% for Plaque Psoriasis.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC08
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ilumya (Experimental): Ilumya 100mg subcutaneous at weeks 0, 4 and 16.
  Interventions: Drug: Ilumya Injectable Product

INTERVENTIONS:
Drug: Ilumya Injectable Product — IL-23 injection

SUMMARY:
Patient with moderate-to-severe plaque psoriasis will receive Ilumya with or without Halog ointment.

DETAILED DESCRIPTION:
25 adult subjects with moderate to severe plaque psoriasis will receive Ilumya 100mg subcutaneously at weeks 0, 4 and 16.

At week 16, patients with remaining BSA ˃3% will be given HALOG ointment 0.1% to apply BID for 4 weeks. Patients who have ≤3% BSA at week 16 will remain on Ilumya monotherapy.

Patients will continue to be evaluated at weeks 20 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age;
2. Diagnosis of moderate-to-severe chronic plaque-type psoriasis as defined by

   * BSA 10%
   * PGA ≥3
   * PASI ≥12
3. Must be a candidate for phototherapy and/or systemic therapy
4. Females of childbearing potential (FCBP) must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.

Exclusion Criteria:

1. Non-plaque forms of psoriasis
2. Women of childbearing potential who are pregnant, intend to become pregnant, or are lactating
3. Presence of significant uncontrolled medical condition that in the opinion of the investigator would affect patient safety during the trial.
4. Active or untreated latent tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Body surface area | 16 weeks
  evaluation of body surface area percentage affected by psoriasis where 1 palm is equivalent to 1%

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No